CLINICAL TRIAL: NCT05342376
Title: Role of Dexmeditomidine HCL for Prevention of Shivering in Obstetrical Spinal Anesthesia, a Randomized Controlled Double Blind Parallel Study.
Brief Title: Intravenous Dexmeditomidine for Prevention of Spinal Anesthesia Induced Shivering.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Mohammad Shafiq, Consultant Anesthesiologist, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RMI/RMI-REC/Approval/58
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Shivering; Cesarean Delivery
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The study design is prospective double-blinded randomized controlled parallel trial with allocation ratio of 1:1.
Who Masked: Participant, Care Provider
Masking Description: Two color coded envelops containing drug and placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): This is group D, which will receive 10 micro-gram Dexmeditomidine diluted in 02 ml normal saline to be administered intravenously in 10 minutes after umbilical cord is clamped..
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Saline (Active Comparator): This group S will receive 02 ml normal saline intravenously as placebo in 10 minutes after umbilical cord is clamped..
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — The parturients will receive 10 micro-gram Dexmedetomidine diluted in 02 ml normal saline to be administered intravenously over 10 minutes after umbilical cord is clamped..
  Other Names: inj Precidex (brookes pharmaceutical, Pakistan)
  Arms: Dexmedetomidine
Drug: Normal Saline — The parturients will receive 02 ml normal saline as placebo, to be administered intravenously over 10 minutes after umbilical cord is clamped.
  Other Names: Normal Saline 0.9 %
  Arms: Saline

SUMMARY:
Intraoperative and post operative shivering is a common problem encountered in operating rooms and recovery suites. Shivering under spinal anesthesia has an incidence of 40-60%. Shivering is not only uncomfortable for the patient; additionally it increases minute oxygen consumption, subjecting the patient to a higher risk of cardiovascular complications. A variety of drugs like pethidine, fentanyl, alfentanil, sufentanil, buprenorphine, doxapram, clonidine, and ketanserin, are reported to be effective in suppressing postoperative shivering, yet an ideal drug/ method to be explored. Dexmeditomidine, a sedative and analgesic, may control shivering without significant adverse effects, like nausea and vomitting and respiratory depression.

The study design will be randomized controlled parallel trials with sample size of 80,They will be randomized into two equal groups. One group will receive 10 microgram Inj. Dexmeditomedine while the other will recieve inj. normal saline as placebo. The participants will be assessed for intra- and postoperative shivering.

DETAILED DESCRIPTION:
Intraoperative inadvertent changes in the body temperature are quite common. Incidence of inadvertent hypothermia (up to 90%) is much higher than hyperthermia. The hypothermic patients shiver postoperatively after general anesthesia and both introperatively and post operatively during regional anesthesia. Shivering under spinal anesthesia has an incidence of 40-60%. Shivering is not only uncomfortable for the patient; additionally it increases minute oxygen consumption VO2 at the cost of increased presser hormones level, subjecting the patient to a higher risk of cardiovascular complications. Heat loss from skin and surgical site is mostly by radiation. Dropped body temperature in cesarean section under spinal anesthesia is due to a combination of anesthetic-induced impaired thermoregulation i.e. vasodilation and inhibition of vasoconstriction in the blocked dermatomes, which are due to autonomic and motor blockade caused by spinal anesthesia. General anesthesia also leads to hypothermia due to vasodilation and reduced metabolic rate, in the order of 20%-30%. Additional factors are exposure to cold environment, un-warmed cold irrigants/ intra vascular fluids and ventilation with dry anesthetic gases. In spinal anesthesia, due to blocked motor activity below umbilicus, shivering in response to hypothermia is abolished. It interferes with physiologic heat recovery, as human core body temperature should normally be maintained within the narrow range of 36.5-37.5 °C. A variety of drugs like pethidine, fentanyl, alfentanil, sufentanil, buprenorphine, doxapram, clonidine, and ketanserin, are reported to be effective in suppressing postoperative shivering, yet an ideal drug/ method to be explored. Dexmeditomidine which is an alpha-2 agonist, is a new drug used for analgesia and sedation either in perioperative settings or in intensive care units. It is 7-8 times selective alpha 2 agonist than clonidine and was expected to control shivering like clonidine. There are study demonstrating the favorable effect of Dexmeditomidine via infusion in the intraoperative period on shivering after abdominal hysterectomy. In previous studies, a prophylactic single dose of Dexmeditomidine for prevention or aborting shivering was generally found to be effective after general or regional anesthesia. Dexmedetomidine 0.5 mcg/kg I/v as loading dose was found 100% effective in managing post anesthesia shivering after general anesthesia in children. In another study, it was observed that Dexmedetomidine was equally effective compared to tramadol, and was associated with shorter time for complete shivering control and less incidence of nausea vomiting, but prospects of a single sub loading dose in parturients during spinal anesthesia requires exploration as physiologic volume loaded parturients at term are expected to lose more heat by redistribution due to vasodilation caused by spinal anesthesia.

OBJECTIVE: To determine the role of single sub loading dose of Dexmeditomidine i.e. 10 mcg (0.1- 0.2 microgram/kg) administered intravenously for prevention of shivering in participants undergoing Cesarean section under spinal anesthesia in a randomized double-blind, placebo controlled parallel study.

ELIGIBILITY:
Inclusion criteria:

* American Society of Anesthesiologists (ASA) physical status I and II ladies
* Singleton pregnancies.
* Undergoing elective Cesarean delivery under spinal anesthesia.
* Systolic blood pressure ≥ 100 mm of Hg after umbilical cord clamping

Exclusion criteria:

* ASA class III or above
* Hyperthyroidism
* Cardiopulmonary or respiratory disease
* A psychological disorder
* An initial body temperature of >37.5 °C or <36.5 °C
* Systolic blood pressure <100 mm of Hg after umbilical cord clamping and/or mean arterial pressure (MAP) < 65 mm of Hg after umbilical cord clamping

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Childbearing female, parturients presenting for Cesarean delivery.
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of shivering in all parturients who received either Dexmeditomidine HCL or placebo | Two hours
  The intensity of postoperative shivering will be graded using Bedside Shivering Assessment Scale(BSAS) from 0 - 3 with 0= no shivering and 3=severe shivering.

SECONDARY OUTCOMES:
Rate of sedation in all parturients who received either Dexmedetomidine HCL or placebo. | Two hours
  Sedation will be assessed through Richmond agitation sedation scale (RASS) from +4 to - 5 with +4= combative and -5= unarousable.
Rate of postoperative pain and analgesia in all parturients who received either Dexmeditomidine HCL or placebo. | Two hours
  Postoperative pain/analgesia will be assessed through visual analogue scale (VAS) with 0= no pain, 100= very severe pain.
Incidence of adverse reactions associated with Dexmedetomidine HCL | Two hours
  Incidence of adverse reactions like hypotension and bradycardia in Dexmedetomidine group will be noted and compared with saline group

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shafiq, FCPS, Principal Investigator — Rehman Medical Institute
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Yes Data including clinical and demographic characteristics, not affecting patient's confidentiality, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April, 2022 to April, 2025
Access Criteria: IPD will be shared on inter institutional request basis.

REFERENCES:
- [Background] 2. Bhattacharya P, Bhattacharya L, Jain RK, Agarwal RC (2003) Postanaesthesia shivering (PAS): A review. Indian J Anaesth 47: 88-93.
- [Background] Buggy DJ, Crossley AW. Thermoregulation, mild perioperative hypothermia and postanaesthetic shivering. Br J Anaesth. 2000 May;84(5):615-28. doi: 10.1093/bja/84.5.615. No abstract available. PMID 10844839
- [Background] Bindu B, Bindra A, Rath G. Temperature management under general anesthesia: Compulsion or option. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):306-316. doi: 10.4103/joacp.JOACP_334_16. PMID 29109627
- [Background] Robinson BJ, Ebert TJ, O'Brien TJ, Colinco MD, Muzi M. Mechanisms whereby propofol mediates peripheral vasodilation in humans. Sympathoinhibition or direct vascular relaxation? Anesthesiology. 1997 Jan;86(1):64-72. doi: 10.1097/00000542-199701000-00010. PMID 9009941
- [Background] Stevens WC, Cromwell TH, Halsey MJ, Eger EI 2nd, Shakespeare TF, Bahlman SH. The cardiovascular effects of a new inhalation anesthetic, Forane, in human volunteers at constant arterial carbon dioxide tension. Anesthesiology. 1971 Jul;35(1):8-16. doi: 10.1097/00000542-197107000-00005. No abstract available. PMID 4932622
- [Background] Piper SN, Suttner SW, Schmidt CC, Maleck WH, Kumle B, Boldt J. Nefopam and clonidine in the prevention of postanaesthetic shivering. Anaesthesia. 1999 Jul;54(7):695-9. doi: 10.1046/j.1365-2044.1999.00849.x. PMID 10417466 (Retraction: PMID 21826813 Anaesthesia. 2011 Jul;66(7):647)
- [Background] Terasako K, Yamamoto M. Comparison between pentazocine, pethidine and placebo in the treatment of post-anesthetic shivering. Acta Anaesthesiol Scand. 2000 Mar;44(3):311-2. doi: 10.1034/j.1399-6576.2000.440316.x. PMID 10714846
- [Background] Iwakiri H, Oda Y, Asada A, Ozaki M. The efficacy of continuous infusion of low dose dexmedetomidine for postoperative patients recovering in general wards. Eur J Anaesthesiol. 2012 May;29(5):251-4. doi: 10.1097/EJA.0b013e3283529ba8. No abstract available. PMID 22450531
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Elvan EG, Oc B, Uzun S, Karabulut E, Coskun F, Aypar U. Dexmedetomidine and postoperative shivering in patients undergoing elective abdominal hysterectomy. Eur J Anaesthesiol. 2008 May;25(5):357-64. doi: 10.1017/S0265021507003110. Epub 2008 Jan 21. PMID 18205960
- [Background] Usta B, Gozdemir M, Demircioglu RI, Muslu B, Sert H, Yaldiz A. Dexmedetomidine for the prevention of shivering during spinal anesthesia. Clinics (Sao Paulo). 2011;66(7):1187-91. doi: 10.1590/s1807-59322011000700011. PMID 21876972
- [Background] Günaydın B, Özköse Z, Tarhan B. Intravenous dexmedetomidine sedation for spinal anesthesia in the prone knee-chest position for lumbar laminectomy surgery. Turk J Med Sci 2004; 34: 353-5.
- [Background] Mittal G, Gupta K, Katyal S, Kaushal S. Randomised double-blind comparative study of dexmedetomidine and tramadol for post-spinal anaesthesia shivering. Indian J Anaesth. 2014 May;58(3):257-62. doi: 10.4103/0019-5049.135031. PMID 25024466
- [Background] Blaine Easley R, Brady KM, Tobias JD. Dexmedetomidine for the treatment of postanesthesia shivering in children. Paediatr Anaesth. 2007 Apr;17(4):341-6. doi: 10.1111/j.1460-9592.2006.02100.x. PMID 17359402
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Result] Moola S, Lockwood C. Effectiveness of strategies for the management and/or prevention of hypothermia within the adult perioperative environment. Int J Evid Based Healthc. 2011 Dec;9(4):337-45. doi: 10.1111/j.1744-1609.2011.00227.x. PMID 22093385